CLINICAL TRIAL: NCT06702709
Title: EFFECTS of INSTRUMENT-ASSISTED SOFT TISSUE MOBILIZATION VS. NEURODEVELOPMENTAL THERAPY on MOTOR FUNCTION in CHILDREN with GMFCS LEVEL I and II SPASTIC DIPLEGIC CEREBRAL PALSY
Brief Title: Comparing the Instrument-Assisted Soft Tissue Mobilization and Neurodevelopmental Therapy for Gross Motor Functions, Muscle Tone and Spasticity in Children with Spastic Diplegic Cerebral Palsy (GMFCS Levels I and II)
Acronym: IASTM;NDT;CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Hamza Ahmed, MPhil Student, Ziauddin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 8211223HAREH
Record Dates: First submitted 2024-11-19; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-03

CONDITIONS: Diplegic Spastic Cerebral Palsy
Keywords: Cerebral Palsy, GMFM, Spasticity
MeSH Terms: conditions — Cerebral palsy, spastic, diplegic; Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): The treatment protocol of the IASTM group will consist on the preparation phase, application phase followed by strengthening. The session is given for 40 minutes for 4 weeks and 3 days per week.
  Interventions: Other: Instrument Assisted Soft Tissue Mobilization
- Group B (Active Comparator): The neurodevelopment therapy for spastic diplegic cerebral palsy includes tone-inhibitory postures. This study will use five-tone inhibitory postures that will be appropriate for the reduction of muscle tone, elongation of lower extremities muscles, and improve gross motor function by enhancing balance and stability. The session is given for 40 minutes for 4 weeks and 3 days per week
  Interventions: Other: Neurodevelopmental Therapy

INTERVENTIONS:
Other: Instrument Assisted Soft Tissue Mobilization — The IASTM method will be applied bilaterally to each target muscle, duration 25 minutes. During treatment, three repetitions are performed on each target muscle, with each repetition lasting 50 seconds. The IASTM technique will be applied at a 60-degree angle. The application sequence follows a specific pattern: For the first 10 seconds, light pressure will be applied during the sweeping stroke, and for the next 20 seconds, moderate pressure will apply during the fanning and brushing strokes. Finally, 10 seconds of deep pressure will administer utilizing oblique sweeping strokes. To help the tissues relax, the treatment will finish with mild sweeping and broad strokes on the hamstring region for 10 seconds
  Other Names: IASTM
  Arms: Group A
Other: Neurodevelopmental Therapy — The neurodevelopment therapy for spastic diplegic cerebral palsy includes tone-inhibitory postures. This study will use five-tone inhibitory postures that will be appropriate for the reduction of muscle tone, elongation of lower extremities muscles, and improve gross motor function by enhancing balance and stability. The following posture will be repeated 3 times on the bilateral lower limb in one session and maintained for 50 seconds with 60 seconds rest between each posture. The total duration of NDT will be 25 minutes.
  Other Names: NDT
  Arms: Group B

SUMMARY:
Cerebral palsy is a neurological condition that affects individuals worldwide, with a global burden of 0.9%. However, prevalence rates show regional variation, with high-income countries reporting rates of 0.2% and low-income countries of 0.3%. In Pakistan, cerebral palsy is the third most common (10.5%) neurological condition in the child population, with a significantly higher frequency of 1.22 per 1000 live births. Amongst the various subtypes of cerebral palsy, spastic diplegic cerebral palsy and spastic quadriplegic cerebral palsy are the most prevalent, accounting for 39% of cases, followed by athetoid (3.34%) and ataxic (10.1%) cerebral palsy in Pakistan.

Individuals with spastic diplegic cerebral palsy exhibit distinct characteristics, including increased muscle tone, scissoring of the lower extremities, and functional impairment. Scissors in the lower limbs, a common manifestation in spastic diplegic cerebral palsy, often result from of hamstring and gastrocnemius hypertonia. The modified Ashworth scale is a sensitive and reliable tool commonly used to assess hypertonicity. This condition primarily results from spasticity caused by upper motor neuron lesions, resulting in excessive alpha motor neuron activity that increases the stretch reflex and muscle tone. Fortunately, spastic diplegic cerebral palsy can be managed with various pharmacological and non-pharmacological approaches.

Pharmacological management includes the use of oral baclofen and botulinum toxin injections. Surgical interventions such as intrathecal baclofen and muscle lengthening procedures are also used to reduce spasticity. However, physical therapy plays a vital role in the management of spastic diplegic cerebral palsy and is critical to improving outcomes for affected individuals. Various physical therapy approaches have been used effectively, including neurodevelopmental therapies, strengthening, passive stretching, strength training combined with stretching, restriction-induced movement therapy and targeted motor reduction programs. Despite their effectiveness, these methods have inherent limitations, such as the limited range of motion with the balance ball, the long time required for motion limitation therapy, and the discomfort associated with stretching exercises. Additionally, differences in practices between therapists were observed.

To address these limitations and improve therapeutic outcomes, the concept of "Instrument Assisted Soft Tissue Mobilization (IASTM)" was introduced. IASTM is a skilled technique involving the use of specialized tools to manipulate the skin, myofascia, muscles, and tendons using direct compression stroke techniques. The application of IASTM tools helps release soft tissue with myofascial adhesions, leading to pain relief, improved range of motion, and improved function. In the context of cerebral palsy, the IASTM is a promising approach, affecting two-point discrimination, pressure pain threshold, and local temperature. In addition, IASTM can promote connective tissue remodeling by breaking down scar tissue, adhesions, and fascial restrictions. In addition, it has been shown to reduce muscle tone by stimulating mechanoreceptors that activate inhibitory interneurons in the spinal cord, leading to decreased activity of alpha motor neurons in extrafusal fibers.

Despite evidence supporting the beneficial impact of IASTM on the special needs population, there is still a paucity of literature on the use of IASTM tools and their effects, particularly for individuals with cerebral palsy. To the best of our knowledge, the use of IASTM is a novel therapeutic approach in the cerebral palsy population of Pakistan to manage muscle tone, range of motion of knee extension and ankle dorsiflexion, and gross motor function. Therefore, this study aims to explore the potential benefits of IASTM in this specific population and aims to provide valuable insights for future research and therapeutic interventions.

DETAILED DESCRIPTION:
A total of 60 participants were recruited for this study after obtaining informed, voluntary assent from the guardians of the participants. Each participant was randomly allocated to group A (n=30), which received Instrument Assisted Soft Tissue Mobilization (IASTM), or group B (n=30), which received neurodevelopmental therapy (NDT). Moreover, the envelope method of simple random sampling was used for group allocation, ensuring that the participants remained blind to their group assignment.

Each participant underwent a baseline assessment before starting the intervention, which lasted 4 weeks. After the 4-week intervention period, the interventions were stopped while standard physical therapy continued, and participants were assessed to measure the immediate effects of both IASTM and neurodevelopmental therapy. Subsequently, a follow-up assessment was carried out at week 8 to evaluate any residual effects of the interventions.

During the study, three participants from the IASTM group and eight participants from the NDT group dropped out, resulting in final groups of 27 participants in group A and 22 participants in group B, respectively. The outcome measures included the Modified Ashworth Scale for hypertonicity assessment, the Universal Goniometer for range of motion (ROM) of knee extension and ankle dorsiflexion, and dimensions D and E of GMFM-88 for evaluating gross motor skills.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with diagnosed Diplagic cerebral palsy are referred by a physician
* Age 4-12 years.
* Children with mild to moderate spasticity according to the Modified Ashworth scale (grade 1, 1+).
* Children with GMFCS level-I and II will be included.
* Children with pseudomyostatic contractures

Exclusion Criteria:

* Localized infectious disease.
* Inflammatory skin condition.
* Diagnosed soft tissue injury of hamstring/gastrocnemius.
* Open wound.
* Osteomyelitis
* Children with a history of any lower limb surgical intervention.
* Sensory impairments especially in lower extremities.
* History of botulinum toxin injections within 4 months before study entry .

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth scale | Baseline
  The Modified Ashworth Scale is a clinical tool developed to assess muscle tone in people with neurological conditions such as cerebral palsy, spinal cord injury, or stroke.The scale rates muscle tone from 0 to 4, with 0 denoting no increase in muscle tone and 4 denoting affected part is rigid in flexion or extension. In this study the modified ashworth scale give the quantitative evaluation of hamstring and gastrocnemius muscle.
Modified Ashworth scale | 4 Week
  The Modified Ashworth Scale is a clinical tool developed to assess muscle tone in people with neurological conditions such as cerebral palsy, spinal cord injury, or stroke.The scale rates muscle tone from 0 to 4, with 0 denoting no increase in muscle tone and 4 denoting affected part is rigid in flexion or extension. In this study the modified ashworth scale give the quantitative evaluation of hamstring and gastrocnemius muscle.
Modified Ashworth scale | 8 Week
  The Modified Ashworth Scale is a clinical tool developed to assess muscle tone in people with neurological conditions such as cerebral palsy, spinal cord injury, or stroke.The scale rates muscle tone from 0 to 4, with 0 denoting no increase in muscle tone and 4 denoting affected part is rigid in flexion or extension. In this study the modified ashworth scale give the quantitative evaluation of hamstring and gastrocnemius muscle.
Universal Goniometer | Baseline
  A universal goniometer is a gadget that is used to precisely measure joint angles and range of motion. Typically, it has two moveable arms, such as rulers, that can be adjusted to accommodate various body regions and angles. This study evaluate the range of motion of Knee extension and ankle dorsiflexion.
Universal Goniometer | 4 Week
  A universal goniometer is a gadget that is used to precisely measure joint angles and range of motion. Typically, it has two moveable arms, such as rulers, that can be adjusted to accommodate various body regions and angles. This study evaluate the range of motion of Knee extension and ankle dorsiflexion.
Universal Goniometer | 8 Week
  A universal goniometer is a gadget that is used to precisely measure joint angles and range of motion. Typically, it has two moveable arms, such as rulers, that can be adjusted to accommodate various body regions and angles. This study evaluate the range of motion of Knee extension and ankle dorsiflexion.
Gross Motor Function Measure-88 | Baseline
  Gross Motor Function Measure-88 (GMFM-88), a widely accepted clinical assessment tool, has been developed to evaluate and assess gross motor function in children with cerebral palsy. GMFM-88 evaluate a child's ability to perform a variety of gross motor skills, such as lying and rolling, sitting, crawling and kneeling, standing, walking, running, and jumping. It consists of 88 items that are categorized into five dimensions. In this study the author will be going to use walking, running, and jumping that is dimension E.
Gross Motor Function Measure-88 | 4 Week
  Gross Motor Function Measure-88 (GMFM-88), a widely accepted clinical assessment tool, has been developed to evaluate and assess gross motor function in children with cerebral palsy. GMFM-88 evaluate a child's ability to perform a variety of gross motor skills, such as lying and rolling, sitting, crawling and kneeling, standing, walking, running, and jumping. It consists of 88 items that are categorized into five dimensions. In this study the author will be going to use walking, running, and jumping that is dimension E.
Gross Motor Function Measure-88 | 8 Week
  Gross Motor Function Measure-88 (GMFM-88), a widely accepted clinical assessment tool, has been developed to evaluate and assess gross motor function in children with cerebral palsy. GMFM-88 evaluate a child's ability to perform a variety of gross motor skills, such as lying and rolling, sitting, crawling and kneeling, standing, walking, running, and jumping. It consists of 88 items that are categorized into five dimensions. In this study the author will be going to use walking, running, and jumping that is dimension E.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Abid Khan, Study Chair — Ziauddin University
Locations (1):
- Ziauddin College of Physical Therapy, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramey SL, DeLuca SC, Stevenson RD, Conaway M, Darragh AR, Lo W; CHAMP. Constraint-Induced Movement Therapy for Cerebral Palsy: A Randomized Trial. Pediatrics. 2021 Nov;148(5):e2020033878. doi: 10.1542/peds.2020-033878. Epub 2021 Oct 14. PMID 34649982
- [Background] Novak I, Morgan C, Fahey M, Finch-Edmondson M, Galea C, Hines A, Langdon K, Namara MM, Paton MC, Popat H, Shore B, Khamis A, Stanton E, Finemore OP, Tricks A, Te Velde A, Dark L, Morton N, Badawi N. State of the Evidence Traffic Lights 2019: Systematic Review of Interventions for Preventing and Treating Children with Cerebral Palsy. Curr Neurol Neurosci Rep. 2020 Feb 21;20(2):3. doi: 10.1007/s11910-020-1022-z. PMID 32086598
- [Background] Kim J, Sung DJ, Lee J. Therapeutic effectiveness of instrument-assisted soft tissue mobilization for soft tissue injury: mechanisms and practical application. J Exerc Rehabil. 2017 Feb 28;13(1):12-22. doi: 10.12965/jer.1732824.412. eCollection 2017 Feb. PMID 28349028
- [Background] Kalkman BM, Holmes G, Bar-On L, Maganaris CN, Barton GJ, Bass A, Wright DM, Walton R, O'Brien TD. Resistance Training Combined With Stretching Increases Tendon Stiffness and Is More Effective Than Stretching Alone in Children With Cerebral Palsy: A Randomized Controlled Trial. Front Pediatr. 2019 Aug 13;7:333. doi: 10.3389/fped.2019.00333. eCollection 2019. PMID 31456995
- [Background] Kalkman BM, Bar-On L, Cenni F, Maganaris CN, Bass A, Holmes G, Desloovere K, Barton GJ, O'Brien TD. Muscle and tendon lengthening behaviour of the medial gastrocnemius during ankle joint rotation in children with cerebral palsy. Exp Physiol. 2018 Oct;103(10):1367-1376. doi: 10.1113/EP087053. Epub 2018 Sep 13. PMID 30091806
- [Background] Hilderley AJ, Wright FV, Taylor MJ, Chen JL, Fehlings D. Functional Neuroplasticity and Motor Skill Change Following Gross Motor Interventions for Children With Diplegic Cerebral Palsy. Neurorehabil Neural Repair. 2023 Jan;37(1):16-26. doi: 10.1177/15459683221143503. Epub 2022 Dec 15. PMID 36524254
- [Background] Duffy S, Martonick N, Reeves A, Cheatham SW, McGowan C, Baker RT. Clinician Reliability of One-Handed Instrument-Assisted Soft Tissue Mobilization Forces During a Simulated Treatment. J Sport Rehabil. 2022 May 1;31(4):505-510. doi: 10.1123/jsr.2021-0216. Epub 2022 Feb 2. PMID 35108674
- [Background] Tekin F, Kavlak E, Cavlak U, Altug F. Effectiveness of Neuro-Developmental Treatment (Bobath Concept) on postural control and balance in Cerebral Palsied children. J Back Musculoskelet Rehabil. 2018;31(2):397-403. doi: 10.3233/BMR-170813. PMID 29171980
- [Background] Simatou M, Papandreou M, Billis E, Tsekoura M, Mylonas K, Fousekis K. Effects of the Ergon(R) instrument-assisted soft tissue mobilization technique (IASTM), foam rolling, and static stretching application to different parts of the myofascial lateral line on hip joint flexibility. J Phys Ther Sci. 2020 Apr;32(4):288-291. doi: 10.1589/jpts.32.288. Epub 2020 Apr 2. PMID 32273652
- [Background] Sadowska M, Sarecka-Hujar B, Kopyta I. Cerebral Palsy: Current Opinions on Definition, Epidemiology, Risk Factors, Classification and Treatment Options. Neuropsychiatr Dis Treat. 2020 Jun 12;16:1505-1518. doi: 10.2147/NDT.S235165. eCollection 2020. PMID 32606703
- [Background] Rivera-Rujana DM, Munoz-Rodriguez DI, Agudelo-Cifuentes MC. Reliability of the Gross Motor Function Measure-66 scale in the evaluation of children with cerebral palsy: validation for Colombia. Bol Med Hosp Infant Mex. 2022;79(1):33-43. doi: 10.24875/BMHIM.21000094. PMID 35086134
- [Background] O'Sullivan R, Marron A, Brady K. Crouch gait or flexed-knee gait in cerebral palsy: Is there a difference? A systematic review. Gait Posture. 2020 Oct;82:153-160. doi: 10.1016/j.gaitpost.2020.09.001. Epub 2020 Sep 6. PMID 32927222
- [Background] Nahm NJ, Graham HK, Gormley ME Jr, Georgiadis AG. Management of hypertonia in cerebral palsy. Curr Opin Pediatr. 2018 Feb;30(1):57-64. doi: 10.1097/MOP.0000000000000567. PMID 29135566
- [Background] Ayala L, Winter S, Byrne R, Fehlings D, Gehred A, Letzkus L, Noritz G, Paton MCB, Pietruszewski L, Rosenberg N, Tanner K, Vargus-Adams J, Novak I, Maitre NL. Assessments and Interventions for Spasticity in Infants With or at High Risk for Cerebral Palsy: A Systematic Review. Pediatr Neurol. 2021 May;118:72-90. doi: 10.1016/j.pediatrneurol.2020.10.014. Epub 2020 Nov 4. PMID 33563492
- [Background] Yoo M, Ahn JH, Rha DW, Park ES. Reliability of the Modified Ashworth and Modified Tardieu Scales with Standardized Movement Speeds in Children with Spastic Cerebral Palsy. Children (Basel). 2022 Jun 3;9(6):827. doi: 10.3390/children9060827. PMID 35740764
- [Background] Rafique A, Naz H. A survey-based report on the occurrence of cerebral palsy in Urban areas of Karachi. J Pak Med Assoc. 2020 Aug;70(8):1442-1444. doi: 10.5455/JPMA.28135. PMID 32794503
- [Background] Chand P, Sultan T, Kulsoom S, Jan F, Ibrahim S, Mukhtiar K, Awan S, Rafique I, Khan DSA, Sulaiman A, Saqib MAN, Sajid M, Padhani ZA, Das JK, Soomro S, Wasay M. Spectrum of Common Pediatric Neurological Disorders: A Cross-Sectional Study From Three Tertiary Care Centres Across Pakistan. Pediatr Neurol. 2023 Jan;138:33-37. doi: 10.1016/j.pediatrneurol.2022.09.005. Epub 2022 Oct 7. PMID 36335840
- [Background] McIntyre S, Goldsmith S, Webb A, Ehlinger V, Hollung SJ, McConnell K, Arnaud C, Smithers-Sheedy H, Oskoui M, Khandaker G, Himmelmann K; Global CP Prevalence Group*. Global prevalence of cerebral palsy: A systematic analysis. Dev Med Child Neurol. 2022 Dec;64(12):1494-1506. doi: 10.1111/dmcn.15346. Epub 2022 Aug 11. PMID 35952356
- [Background] Olusanya BO, Smythe T, Ogbo FA, Nair MKC, Scher M, Davis AC. Global prevalence of developmental disabilities in children and adolescents: A systematic umbrella review. Front Public Health. 2023 Feb 16;11:1122009. doi: 10.3389/fpubh.2023.1122009. eCollection 2023. PMID 36891340
- See also: Related Info — https://www.kmuj.kmu.edu.pk/article/view/16033
- See also: Related Info — https://www.gup.ugal.ro/ugaljournals/index.php/efms/article/view/4432